CLINICAL TRIAL: NCT03313492
Title: Modifying Young Adult Skin Cancer Risk and Protective Behaviors (UV4.me2): A Hybrid Type 2 Dissemination/Effectiveness Trial
Brief Title: Modifying Young Adult Skin Cancer Risk and Protective Behaviors
Acronym: UV4me2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: University of Pennsylvania (Other); ITX Corporation (Unknown); RTI International (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Dr. Carolyn Heckman, Ph.D, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro2018001543; R01CA204271 (NIH)
Record Dates: First submitted 2017-10-04; First posted 2017-10-18 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Melanoma and Other Malignant Neoplasms of Skin
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- E-Pamphlet (Active Comparator): A free non-interactive e-pamphlet ("Skin Cancer Prevention and Early Detection" from the American Cancer Society) will be accessible via our website.
  Interventions: Behavioral: E-Pamphlet
- Original UV4.me (Active Comparator): Participants will view the original UV4.me web intervention, which includes educational modules, personalized responses to quizzes, information on skin type and burn risk, UV damage photo of similar individuals, avatar activity, age progression images, personal risk calculator, SPF (sun protection factor) calculator. The website content will remain the same, with the exception of updating photos, statistics, and cultural references for the current year.
  Interventions: Behavioral: UV4.me
- Enhanced UV4.me2 (Experimental): Participants will view an enhanced version of the UV4.me website. Improvements to the website are based on user feedback from the original UV4.me trial, as well as reviews and models of effective e-Health interventions and implementation strategies.
  Interventions: Behavioral: UV4.me2

INTERVENTIONS:
Behavioral: UV4.me2 — UV4.me2 is an enhanced version of the original UV4.me web intervention and features the many of the same educational material and interactive components. New features/strategies for reach, effectiveness, and implementation include:
  1. A mobile version of the site
  2. Incentives in the form of clickable coupons and links to free samples for sun protection products (e.g., sunscreen)
  3. Behavioral tracking and feedback, where users can set goals, track their progress, and receive tailored feedback
  Arms: Enhanced UV4.me2
Behavioral: UV4.me — Original version of the UV4.me website, which offers education and tailored responses to interactive quizzes about current sun protective behaviors and barriers to engaging in sun protective behaviors.
  Arms: Original UV4.me
Behavioral: E-Pamphlet — A free non-interactive e-pamphlet ("Skin Cancer Prevention and Early Detection" from the American Cancer Society). Includes information on skin cancer risk and prevention.
  Arms: E-Pamphlet

SUMMARY:
Skin cancer is the most common cancer and can be deadly, debilitating, damaging, and disfiguring, yet is highly preventable. In 2014, the US Surgeon General made a call to action about the "major public health problem" of skin cancer, noting potential contributions of behavioral science and education, and a need for investments in such efforts. Almost five million Americans are treated for skin cancer annually, and incidence is rising. Risk factors for melanoma and non-melanoma skin cancers include personal or family history of skin cancer, certain physical characteristics (e.g., fair skin, numerous moles), as well as excessive ultraviolet (UV) radiation exposure. Our work shows that skin cancer risk behaviors, including sunburns, indoor tanning, and lack of protection peak at age 25. Thus, young adulthood is an important window for skin cancer risk reduction interventions. However, young adults tend to be resistant to public health recommendations because, as a group, they perceive themselves as having more immediate priorities than disease prevention, that the consequences of their current health behaviors are in the distant future, and they also tend to be experimenters and risk-takers highly influenced by peers.

The principal investigator developed a web-based intervention (UV4.me) that was found to significantly decrease UV exposure and increase skin protection behaviors among young adults in a randomized controlled trial of nearly 1000 participants.

The objective of this project is to investigate the reach, effectiveness, implementation, maintenance, and cost of an enhanced version of that web intervention (UV4.me2) in a large national randomized controlled trial. The ultimate goal is to improve the skin cancer protection behaviors (and potentially decrease skin cancer incidence) among a national sample of young adults at moderate to high risk of developing skin cancer.

Primary Aim 1. To enhance and determine intervention reach (i.e., enrollment, representativeness).

Primary Aim 2. To determine the effectiveness of the enhanced intervention.

Secondary Aim 1. To determine maintenance of the UV4.m4 and UV4.me2 interventions through evaluation at 6 and 12-month follow-up.

Secondary Aim 2. To determine intervention implementation by young adults.

Secondary Aim 3. To determine the costs of the UV4.me and UV4.me2 interventions.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to high risk for skin cancer

Exclusion Criteria:

* Not able to speak English
* Past history of skin cancer

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1746 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Reach: eligibility by recruitment source. | 18 months
  The number of participants who are eligible for the study by recruitment source (i.e., skin protection organizations, Google Adwords, Facebook ads, consumer research panel, word of mouth).
Efficacy: Sun protection behaviors | Change from baseline to 3 months
  Skin cancer-related behavioral outcomes will initially be assessed at baseline and 3 months later. Sun protection will be measured using a self-report scale assessing behaviors such as sunscreen use and shade seeking.
Efficacy: UV exposure behaviors | Change from baseline to 3 months
  Skin cancer-related behavioral outcomes will initially be assessed at baseline and 3 months later. UV exposure will be measured using a self-report scale assessing how many times in the past month the subject engaged in behaviors such as sunbathing and using a tanning bed/booth.
Reach: enrollment by recruitment source. | 18 months
  The number of participants who enroll in the study by recruitment source (i.e., skin protection organizations, Google Adwords, Facebook ads, consumer research panel, word of mouth).

SECONDARY OUTCOMES:
Maintenance of skin cancer-related behavioral outcomes (sun protection) | 6 months
  Sun protection behaviors will be assessed at 6 months using a self-report scale assessing behaviors such as sunscreen use and shade seeking.
Maintenance of skin cancer-related behavioral outcomes (sun protection) | 12 months
  Sun protection behaviors will be assessed at 12 months using a self-report scale assessing behaviors such as sunscreen use and shade seeking.
Maintenance of skin cancer-related behavioral outcomes (UV exposure) | 6 months
  UV exposure will be assessed at 6 months using a self-report scale assessing how many times in the past month the subject engaged in behaviors such as sunbathing and using a tanning bed/booth.
Maintenance of skin cancer-related behavioral outcomes (UV exposure) | 12 months
  UV exposure will be assessed at 12 months using a self-report scale assessing how many times in the past month the subject engaged in behaviors such as sunbathing and using a tanning bed/booth.
Implementation: Web intervention use frequency | 1 month
  How frequently participants logged into the interventions will be recorded.
Cost of interventions | Through study completion
  Total costs of the interventions will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Heckman, PhD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (2):
- United States (2):
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heckman CJ, Handorf EA, Darlow SD, Ritterband LM, Manne SL. An online skin cancer risk-reduction intervention for young adults: Mechanisms of effects. Health Psychol. 2017 Mar;36(3):215-225. doi: 10.1037/hea0000420. Epub 2016 Nov 7. PMID 27819460
- [Background] Heckman CJ, Darlow SD, Ritterband LM, Handorf EA, Manne SL. Efficacy of an Intervention to Alter Skin Cancer Risk Behaviors in Young Adults. Am J Prev Med. 2016 Jul;51(1):1-11. doi: 10.1016/j.amepre.2015.11.008. Epub 2016 Jan 22. PMID 26810358
- [Background] Heckman CJ, Handorf E, Darlow SD, Yaroch AL, Raivitch S. Refinement of measures to assess psychosocial constructs associated with skin cancer risk and protective behaviors of young adults. J Behav Med. 2017 Aug;40(4):574-582. doi: 10.1007/s10865-017-9825-3. Epub 2017 Feb 2. PMID 28155000
- [Background] Heckman CJ, Riley M, Khavjou O, Ohman-Strickland P, Manne SL, Yaroch AL, Bhurosy T, Coups EJ, Glanz K. Cost, reach, and representativeness of recruitment efforts for an online skin cancer risk reduction intervention trial for young adults. Transl Behav Med. 2021 Oct 23;11(10):1875-1884. doi: 10.1093/tbm/ibab047. PMID 34160622
- [Derived] Heckman CJ, Mitarotondo A, Lin Y, Khavjou O, Riley M, Manne SL, Yaroch AL, Niu Z, Glanz K. Digital Interventions to Modify Skin Cancer Risk Behaviors in a National Sample of Young Adults: Randomized Controlled Trial. J Med Internet Res. 2024 Jul 2;26:e55831. doi: 10.2196/55831. PMID 38954433

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-07-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT03313492/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/92/NCT03313492/ICF_001.pdf